CLINICAL TRIAL: NCT01222377
Title: Endoscopic Breast Surgery Feasibility Study
Brief Title: Endoscopic Breast Surgery in Treating Patients With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: P.I. left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-09-14; NCI-2010-02088
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo endoscopic breast surgery.
  Interventions: Procedure: endoscopic surgery; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: endoscopic surgery — Undergo endoscopic breast surgery
  Other Names: surgery, endoscopic
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
RATIONALE: Endoscopic breast surgery (EBS) is a less invasive type of surgery for breast cancer and may have fewer side effects and improve recovery. PURPOSE: This clinical trial studies endoscopic breast surgery in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the surgical complication rate in patients undergoing EBS for benign or malignant disease and the 5-year local recurrence rate following endoscopic breast surgery among subjects undergoing EBS for breast cancer at USC. SECONDARY OBJECTIVES: I. To evaluate the safety, breast cosmesis and patient quality of life following EBS. OUTLINE: Patients undergo endoscopic breast surgery. After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer or prophylactic mastectomy requiring axillary nodal staging
* Breast disease (e.g., fibroadenoma, ADH)
* Ability to read and/or comprehend consent form and questionnaires
* Ability to follow-up per protocol
* Not pregnant or breastfeeding

Exclusion Criteria:

* Pregnant or breastfeeding
* Evidence of chest wall or skin* involvement
* NOTE: *may be endoscopy-assisted

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To estimate the surgical complication rate among all patients having EBS and the local recurrence rate among patients with breast cancer | 5 years

SECONDARY OUTCOMES:
To evaluate the safety, breast cosmesis and patient quality of life following EBS | After completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Holmes, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States